CLINICAL TRIAL: NCT04622878
Title: Combined Treatment ( Image Guided Thrombectomy and Endovascular Therapy With Open Femoral Access ) for Acute Limb Ischemia
Brief Title: Combined Management in ALI ( Image Guided Thrombectomy With Open Transfemoral Access )
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kerolos Raafat Khalil Gad, Resident physician at vascular surgery department ، Assiut University, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Combined Management in ALI
Record Dates: First submitted 2020-09-27; First posted 2020-11-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Limb Ischemia
MeSH Terms: interventions — Thrombectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- acute lower limb ischemia patients (Other): patients with no palpable pulsations or audible signals in the lower limb
  Interventions: Procedure: thrombectomy and PTA

INTERVENTIONS:
Procedure: thrombectomy and PTA — open femoral access with fogarty catheter then PTA with balloon and possible stenting if needed

SUMMARY:
Acute limb ischemia (ALI) is a sudden decrease in limb perfusion due to either an embolic or a thrombotic vascular occlusion, defined as the presence of symptoms within two weeks of onset. The profound ischemia represents an emergency in which delayed treatment results in limb loss and, potentially, death. Therefore, timely diagnosis and proper treatments for ALI are important.

Both surgical thrombectomy and endovascular treatment have benefits and drawbacks. Surgical thrombectomy using Fogarty embolectomy catheter has been the standard therapy because it is rapid and effective in cases of embolic ALI. However, blind surgical thrombectomy can result in poor revascularization or unexpected vascular injury in the presence of underlying arterial atherosclerosis or in the presence of subacute and chronic thrombi. In addition, thrombosis of runoff vessels is difficult to remove.

Endovascular management using catheter-directed thrombolysis (CDT) has emerged as an alternative to surgery. It is less invasive, and does not directly damage the vascular endothelium with the capacity to clear thrombus in the small vessels. However, long treatment duration may worsen the clinical situation. Besides, a thrombus of more than two weeks does not respond well to the thrombolysis, and it is difficult to determine the exact stage of thrombus according to the clinical history. These problems may be minimized by combined treatment, which includes surgical thrombectomy and endovascular treatment.

DETAILED DESCRIPTION:
The aim of our research is to evaluate the effectiveness and safety of combined treatment (surgical thrombectomy and endovascular treatment) for ALI with various clinical considerations

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute onset of lower limb pain with various degrees of movement compromise.
* History of intermittent claudication with a sudden worsening of claudication and pain at rest for less than one month.
* Patients with Duplex or MSCT angiography of the lower limbs showing embolic events on healthy vessels or thrombosis of diseased vessels with or without collateralization.
* Thrombus in a poor location that is difficult to be removed by surgical thrombectomy alone.
* Acute lower limb ischemia due to acute arterial graft occlusion

Exclusion Criteria:

* - Medically compromised patients, not fit for the intervention.
* Patients with critical chronic limb ischemia (grade III, IV).
* Patients with known vasculitis or lab investigations suggesting vasculitis before treating the cause.
* Patients who refused the intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
limb salvage | immediately post operative
  Technical success rates is defined as patency of the treated vessel segment with less than 20 % residual stenosis , without dissection and restoration of in line flow to foot , weight and height of the pt will be combined to report BMI kg/m^2

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Kashyap VS, Gilani R, Bena JF, Bannazadeh M, Sarac TP. Endovascular therapy for acute limb ischemia. J Vasc Surg. 2011 Feb;53(2):340-6. doi: 10.1016/j.jvs.2010.08.064. Epub 2010 Nov 3. PMID 21050699